CLINICAL TRIAL: NCT02546479
Title: Breast and Other Cancers Following X-Rays for Scoliosis
Brief Title: Follow-Up Study of People Treated for Scoliosis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Social & Scientific Systems Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915194; 15-C-N194
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07-11

CONDITIONS: Breast and Other Cancer Incidence and Mortality; All Cause Mortality; Circulatory Disease Mortality; Respiratory Disease Mortality
Keywords: Mortality; Radiation; Spine deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patientis: patients diagnosed with scoliosis and other spinal deformities

SUMMARY:
Background:

Scoliosis is a curving of the spine. It usually happens in girls when they are children and teens. Doctors often use x-rays to diagnose it. The x-rays give low radiation. This may increase the risk that those young women get cancer later in life. Researchers want to learn more about this risk. They will look data that has already been collected.

Objectives:

To study cancer risks of repeated low radiation from x-rays for scoliosis. Also, to study death risks related to certain scoliosis patient characteristics. These include causes, kinds of curvature, and kinds of treatment.

Eligibility:

Medical records of women from past scoliosis studies.

Design:

This U.S. Scoliosis Cohort includes more than 5,000 women who were diagnosed between 1912 and 1965.

Data were collected on these women in the 1980s and 1990s. These came from medical records, radiology log books, and x-ray films. Researchers found out where participants were, including if they were dead. Some women were given a follow-up questionnaire.

Researchers want to find out where participants are today. They want to identify new deaths of participants. They want to find out their causes of death. This data will be added to other databases.

DETAILED DESCRIPTION:
U.S. Scoliosis Cohort includes 5,573 female spinal deformity (93% scoliosis) patients diagnosed in any of 14 medical centers in the U.S. during 1912-1965. The primary objective of this study is to evaluate site-specific cancer risks associated with repeated low-dose radiation exposures from diagnostic x-rays. A secondary objective is to evaluate late mortality risks associated with patient characteristics, such as etiology, degree and type of curvature, and type of treatment. The current proposal is to extend mortality follow-up by 10 years. All patients not known to be deceased will be submitted to the National Death Index Plus to identify new deaths and obtain causes of death.

A feasibility study was conducted in four medical centers in the Minneapolis-St. Paul, Minnesota area during 1983-1987. The primary goals of the feasibility study were to ascertain if an adequate number of patients meeting the study criteria could be identified and located, medical and radiography records were available and substantially complete, organspecific radiation doses could be estimated from the available data and were large enough to warrant further study, and a reasonable percentage of patients would complete a follow-up questionnaire. The feasibility study was successful in meeting all goals. Enrolled for study were 1,030 female patients with spinal deformities diagnosed during 1922-1965. Medical records were abstracted, individual x-ray films were reviewed, patients were located, and follow-up questionnaire was administered to identify incident cancers. Eleven breast cancers were reported. Scoliosis patients had an 80% higher breast cancer risk compared to women in the general population and, based on internal cohort analyses, breast cancer risk increased with increasing number of x-rays and with estimated radiation dose to the breast.

An expanded study was conducted during 1988-1993. The main goals of the expanded study were to enlist the collaboration of suitable additional medical centers where large numbers of spinal deformity patients were treated before 1966, abstract data from medical and radiology records, trace patients for vital status and current location, obtain information on incident cancers and cancer risk factors by questionnaire, medically validate reported cancers, and determine causes of death for decedents. Another 4,543 patients diagnosed during 1912-1965 were enrolled from ten hospitals, bringing the total study population to 5,573 patients. Compared to women in the general population, spinal deformity patients had statistically significantly higher risks of dying from breast cancer, and for both incidence and mortality, breast cancer risk increased with increasing diagnostic radiation exposure to the breast. Patients also have elevated risks for mortality from all causes, circulatory, respiratory, nervous system, musculoskeletal, digestive, and infectious & parasitic diseases, primarily related to degree of spinal curvature. Additional mortality follow-up will enable more definitive assessments of cancer and other disease risks with radiation and other factors in these patients.

ELIGIBILITY:
* Data Analysis Only

Ages: 50 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5573 (Actual)
Dates: Start 2015-09-09; Primary Completion 2016-08-16 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Cancer incidence | 1993
  Incidence of breast and other cancers.
Cancer and other disease mortality | 2015
  Mortality from cancer and other causes.

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Doody, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Doody MM, Lonstein JE, Stovall M, Hacker DG, Luckyanov N, Land CE. Breast cancer mortality after diagnostic radiography: findings from the U.S. Scoliosis Cohort Study. Spine (Phila Pa 1976). 2000 Aug 15;25(16):2052-63. doi: 10.1097/00007632-200008150-00009. PMID 10954636
- [Background] Ronckers CM, Doody MM, Lonstein JE, Stovall M, Land CE. Multiple diagnostic X-rays for spine deformities and risk of breast cancer. Cancer Epidemiol Biomarkers Prev. 2008 Mar;17(3):605-13. doi: 10.1158/1055-9965.EPI-07-2628. PMID 18349278
- [Background] Ronckers CM, Land CE, Miller JS, Stovall M, Lonstein JE, Doody MM. Cancer mortality among women frequently exposed to radiographic examinations for spinal disorders. Radiat Res. 2010 Jul;174(1):83-90. doi: 10.1667/RR2022.1. PMID 20681802